CLINICAL TRIAL: NCT00268372
Title: A Phase III Trial of Standard Fractionation Radiation and Concurrent Single Agent Cisplatin, With and Without Docetaxel, Cisplatin, and 5-Fluorouracil Induction Chemotherapy, in Patients With Advanced Oropharyngeal Squamous Cell Cancer
Brief Title: S0427, Combination Chemotherapy & RT in Treating Patients With Stage III or Stage IV Cancer of the Oropharynx
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: SWOG eliminated its head and neck committee
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000459847; S0427 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Docetaxel; Fluorouracil; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cisplatin/RT alone (Active Comparator): cisplatin and radiation therapy
  Interventions: Drug: cisplatin; Radiation: radiation therapy
- induction chemo followed by cisplatin/RT (Experimental): docetaxel, cisplatin and 5-fluorouracil induction chemotherapy followed by surgery and/or cisplatin and radiation therapy
  Interventions: Drug: cisplatin; Drug: docetaxel; Drug: 5-fluorouracil; Procedure: surgery

INTERVENTIONS:
Drug: cisplatin
  Other Names: platinol
Drug: docetaxel
  Other Names: taxotere
  Arms: induction chemo followed by cisplatin/RT
Drug: 5-fluorouracil
  Other Names: 5-FU
  Arms: induction chemo followed by cisplatin/RT
Procedure: surgery
  Arms: induction chemo followed by cisplatin/RT
Radiation: radiation therapy
  Arms: cisplatin/RT alone

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, cisplatin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together with radiation therapy may kill more tumor cells. It is not yet known whether giving combination chemotherapy together with radiation therapy is more effective than giving cisplatin together with radiation therapy in treating cancer of the oropharynx.

PURPOSE: This randomized phase III trial is studying combination chemotherapy and radiation therapy to see how well they work compared to cisplatin and radiation therapy in treating patients with stage III or stage IV cancer of the oropharynx.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with previously untreated stage III or IV squamous cell carcinoma of the oropharynx treated with induction chemotherapy comprising docetaxel, cisplatin, and fluorouracil followed by radiotherapy and cisplatin versus radiotherapy and cisplatin only.
* Compare the progression-free survival in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the quality of life and functional status of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to primary cancer site (base of tongue vs other), nodal extent (N0-1 vs N2-3), radiotherapy plan (conventional [2-D or 3-D conformal radiotherapy] vs intensity modulated radiotherapy). Patients are randomized to 1 of 2 treatment arms.

* Arm I (induction chemotherapy with or without salvage surgery followed by chemoradiotherapy)

  * Induction chemotherapy with or without early salvage surgery: Patients receive docetaxel IV over 1 hour and cisplatin over 30-60 minutes on day 1 and fluorouracil IV continuously on days 1-4. Treatment repeats every 21 days for 1-3 courses. Patients achieving complete or partial response at the primary site after course 1 receive 2 additional courses of therapy and then proceed to chemoradiotherapy within 3-4 weeks after completion of fluorouracil administration. Patients with stable disease or surgically resectable locoregional disease progression undergo early salvage surgery and then proceed to concurrent chemoradiotherapy within 70 days after surgery. Patients with locoregional unresectable disease progression or patients who refused early salvage surgery proceed directly to concurrent chemoradiotherapy within 3-4 weeks after completion of fluorouracil administration.
  * Chemoradiotherapy: Patients undergo 2-D or 3-D conformal radiotherapy or intensity modulated radiotherapy once daily 5 days a week for 7 weeks and receive cisplatin IV over 30-60 minutes concurrently on days 1, 22, and 43* in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients undergoing surgery before chemoradiotherapy receive cisplatin on days 1 and 22 only of a 6-week course of radiotherapy.

* Arm II (chemoradiotherapy only): Patients undergo 2-D or 3-D conformal radiotherapy or intensity modulated radiotherapy once daily 5 days a week for 7 weeks and receive cisplatin IV over 30-60 minutes on days 1, 22, and 43 in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, after completion of chemoradiotherapy, and then at 12 months after randomization.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: Approximately 398 patients (199 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the oropharynx by biopsy or fine needle aspiration of the primary lesion or neck mass

  * Selected stage III or IV disease

    * No T1-2, N1 disease
    * No T4b disease
  * No other primary tumor sites or unknown primary tumor sites
  * Previously untreated disease
* Measurable or non-measurable disease by clinical exam, CT scan or MRI
* Disease considered to be curatively resectable

  * Patients for whom surgical excision is unlikely to result in clear margins are not eligible, including patients with any of the following:

    * Gross extension of tumor to skull base (e.g., T4b disease)
    * Severe trismus
    * Pterygoid plate erosion
    * Sphenoid bone or foramen ovale involvement
    * Direct extension to involve prevertebral-fascia
    * Extension to superior nasopharynx or eustachian tube
    * Direct extension into the neck with involvement of the deep neck musculature (neck node fixation)
    * Suspected invasion (encasement) of the common or internal carotid arteries (T4b)
    * Direct extension of neck disease to involve the external skin
    * Regional metastases to the supraclavicular neck (IVB low level VB nodes)
* Disease must be appropriate for definitive radiotherapy with curative intent
* No evidence of distant metastases (M1)

  * Must have negative chest x-ray

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* No myocardial infarction within the past 3 months
* No unstable or uncontrolled angina
* No active systemic infection
* Granulocyte count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Creatinine < 1.5 mg/dL
* Bilirubin normal
* Alkaline phosphatase ≤ 2 times upper limit of normal (ULN)
* SGOT or SGPT ≤ 1.5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No history of hypersensitivity reaction to products containing polysorbate 80
* No medical contraindication to surgery as defined by the treating institution
* No clinically significant motor or sensory neuropathy ≥ grade 2
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or stage I or II cancer from which the patient is in complete remission

PRIOR CONCURRENT THERAPY:

* No prior therapeutic surgery for head and neck cancer
* No prior radiotherapy
* No prior chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Survival at 2 years | 2 years

SECONDARY OUTCOMES:
Progression-free survival by FACT-HN CTCAE v 3.0 at 2 years | 2 years
Toxicity by CTCAE v 3.0 after induction chemotherapy or after chemotherapy and radiotherapy | after chemotherapy
Incidence of surgical resection | after treatment
Site of relapse | at relapse
Quality of life by FACT-HN week 19 after first and second registration date (arm 1) | after first and second registrations

CONTACTS AND LOCATIONS:
Overall Officials: David J. Adelstein, MD, Study Chair — The Cleveland Clinic; Gregory T. Wolf, MD, Study Director — University of Michigan Rogel Cancer Center; P. G. Shankar Giri, MD, MB, BS, Study Chair — Veterans Affairs Medical Center - Houston
Locations (74):
- United States (74):
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Moline, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Bettendorf, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazooaa, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Capital Health System Regional Cancer Center, Trenton, New Jersey
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - American Fork Hospital, American Fork, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah